CLINICAL TRIAL: NCT04930770
Title: Study About the Response to the Administration of a Third Dose of mRNA-1273 Vaccine (COVID-19 Vaccine Moderna) in Renal Transplants With Immunological Failure Initial to Vaccination
Acronym: VAX-TRES
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No candidates for the trial (all patients have received the third dose of the vaccine)
Sponsor: Maria Joyera Rodríguez (Other)
Responsible Party: Sponsor-Investigator, Maria Joyera Rodríguez, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VAX-TRES; 2021-002356-37 (EudraCT Number)
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Covid19
Keywords: vaccine
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal/renopancreatic transplant's patients with a verified seronegativity (Experimental)
  Interventions: Drug: MRNA-1273

INTERVENTIONS:
Drug: MRNA-1273 — Renal or renopancreatic transplant's patient will receive a third dose of mRNA 1273 (Moderna) vaccine from 28 days after administration of the second dose and after the seronegativity has been verified.

SUMMARY:
The objective will be to analyze the development of cellular and humoral immunity against SARS-CoV-2 after administration of a third dose of mRNA-1273 (Moderna) vaccine in patients who have remained seronegative after the full standard (two-dose) regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Male or female sex;
3. Renal transplant with stable renal function in the last 2 months prior to study inclusion.
4. Had received a full schedule of vaccination for SARS-CoV-2 with mRNA1273 vaccine (Moderna) and remained seronegative at 2 weeks after the second dose.
5. Patient giving written informed consent.

Exclusion Criteria:

1. Renal transplantation < 3 months;
2. Pregnancy or lactation status;
3. Rejection treated within the last 6 months;
4. Presence of humoral immunity to SARS-CoV-2 defined as the presence of specific IgM/IgG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with development of cellular and humoral immunity against SARS-CoV-2 | 2 weeks
  the development of cellular and humoral immunity against SARS-CoV-2 after administration of a third dose of mRNA-1273 (Moderna) vaccine in patients who have remained seronegative after the full standard (two-dose) regimen

SECONDARY OUTCOMES:
Number of patients with development of cellular and humoral immunity against SARS-CoV-2 | 4 months
  development of cellular and humoral immunity against SARS-CoV-2 after 4 months of administration of a third dose of mRNA-1273 vaccine (Moderna).
patient characteristics associated with biological non-response to vaccination | 4 months
  Analysis of baseline factors associated with biological non-response to vaccination, including demographics, comorbidities, and transplant-associated factors. The following items will be reviewed: age, sex, diabetes, type of transplant (kidney-pancreas versus kidney), treatment with anti-thymocyte globulins (ATG) during the last year, lymphopenia defined as < 1000/mm3, time from transplantation < 1 year, eGFR (CKD-EPI), baseline immunosuppression, according to individual drug or the combination received by the patient, type of donor, BMI, ethnicity and blood type.
Incidence of Treatment-Emergent Adverse Events | 4 months
  Percentage of patients with mild and/or severe adverse events after administration of the third dose (safety and tolerability). Number of participants with treatment-related adverse events as assessed by the WHO toxicity scale.